CLINICAL TRIAL: NCT00474851
Title: The Effect of Hormonal Add-Back Therapy in Adolescents Treated With a GnRH Agonist for Endometriosis: A Randomized Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Amy DiVasta, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-01-0004
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Endometriosis
Keywords: Endometriosis; Adolescents; Bone density; GnRH Agonist; Add-back therapy
MeSH Terms: conditions — Endometriosis | interventions — Norethindrone Acetate; Estrogens; Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norethindrone acetate + estrogens (Experimental): Subjects randomized to the experimental arm received add-back therapy with norethindrone acetate 5 mg by mouth daily + conjugated equine estrogens 0.625 mg by mouth daily for the 12 months of study participation.
  Interventions: Drug: Norethindrone acetate + estrogens
- norethindrone acetate + placebo (Placebo Comparator): Subjects randomized to the experimental arm received add-back therapy with norethindrone acetate 5 mg by mouth daily + a placebo capsule by mouth daily for the 12 months of study participation.
  Interventions: Drug: norethindrone acetate + placebo

INTERVENTIONS:
Drug: Norethindrone acetate + estrogens — Norethindrone acetate 5 mg by mouth daily + Conjugated equine estrogens 0.625 mg by mouth daily
  Other Names: Aygestin; Premarin
  Arms: Norethindrone acetate + estrogens
Drug: norethindrone acetate + placebo — norethindrone acetate 5 mg by mouth daily + Placebo capsule 1 pill by mouth daily
  Other Names: Aygestin
  Arms: norethindrone acetate + placebo

SUMMARY:
The purpose of this study is to determine whether a regimen of norethindrone acetate + placebo or norethindrone acetate + conjugated estrogens is superior in maintaining skeletal health and quality of life in adolescents treated with a GnRH agonist for endometriosis.

DETAILED DESCRIPTION:
Endometriosis has become increasingly recognized as a chronic illness which begins during adolescence. Untreated endometriosis may lead to chronic pain and infertility. As recognition of the need for prompt therapy increases, so does the length of time patients will be exposed to treatments. As a result, there exists a pressing need to evaluate adjunctive measures that may limit the associated negative health consequences of treatment.

A gonadotropin-releasing hormone (GnRH) agonist is one medication utilized for patients who have failed other treatments. While GnRH-agonists are effective in relieving symptoms, their long-term use is problematic. GnRH agonists induce a low-estrogen state, causing deleterious effects on bone mineralization. These negative consequences are especially important for our pediatric patients. Adolescence is the critical period in a woman's life for bone acquisition and attainment of peak bone mass. Anything that interferes with this process puts patients at risk for lifelong low bone density and future fracture.

"Add-back" therapy appears to be a promising adjunct to treatment for prevention of this bone loss. Daily therapy with low-doses of hormones preserves bone density in adult patients, without altering the efficacy of the GnRH-agonist. However, no data exist on the effect of add-back therapy in adolescents.

The aim of the current study is to evaluate the safety and efficacy of two add-back regimens, norethindrone acetate + placebo or norethindrone acetate + conjugated estrogens, for the preservation of skeletal health and quality of life in adolescents with endometriosis treated with a GnRH-agonist.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-22 years, at least two years post-menarche
* Body mass index (BMI, kg/m2) between 18 -30 kg/m2
* Surgical diagnosis of endometriosis
* Clinical decision to treat with a GnRH agonist, leuprolide depot (Lupron Depot®; TAP Pharmaceuticals, Inc.) 11.25 mg intra-muscular every 3 months

Exclusion Criteria:

* Concomitant chronic diseases which affect bone health, such as cystic fibrosis, inflammatory bowel disease, renal disease, or diabetes mellitus
* Markedly impaired liver function or liver failure
* Personal history of thromboembolic event (such as deep venous thrombosis)
* Medication use known to affect bone metabolism:

  * Glucocorticoid therapy (including inhaled steroids) or anticonvulsants used in the last 6 months

Ages: 13 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2007-08; Primary Completion 2013-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D DiVasta, MD, MMSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Gallagher JS, DiVasta AD, Vitonis AF, Sarda V, Laufer MR, Missmer SA. The Impact of Endometriosis on Quality of Life in Adolescents. J Adolesc Health. 2018 Dec;63(6):766-772. doi: 10.1016/j.jadohealth.2018.06.027. PMID 30454733
- [Derived] DiVasta AD, Feldman HA, Sadler Gallagher J, Stokes NA, Laufer MR, Hornstein MD, Gordon CM. Hormonal Add-Back Therapy for Females Treated With Gonadotropin-Releasing Hormone Agonist for Endometriosis: A Randomized Controlled Trial. Obstet Gynecol. 2015 Sep;126(3):617-627. doi: 10.1097/AOG.0000000000000964. PMID 26181088

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Conjugated equine estrogens: Conjugated estrogens 0.625 mg PO daily
  Norethindrone acetate: Norethindrone acetate 5 mg PO daily
- Placebo Group: Placebo group
  Placebo: Placebo capsule 1 pill PO daily
  Norethindrone acetate: Norethindrone acetate 5 mg PO daily
Period: Overall Study
Arm/Group | Intervention Group | Placebo Group
Started | 26 | 27
Completed Baseline | 25 | 26
Completed | 18 | 16
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Placebo: Placebo capsule 1 pill PO daily
  Norethindrone acetate: Norethindrone acetate 5 mg PO daily
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.7 (1.4) | 18.1 (1.9) | 17.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: Adjusted mean change in total body areal bone mineral density (aBMD) over the 12 month trial
Time Frame: Baseline to 12 months
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 25 | 26
g/cm^2 | 0.01 (0.006) | -0.11 (0.006)
Statistical Analysis 1: Comparison: Intervention Group vs Placebo Group; Analysis followed the intention-to-treat principle. The time course of each measurement from baseline to 3, 6, 9, and 12 months was compared between arms by repeated-measures analysis of variance (RM-ANOVA), with an autoregressive covariance model to account for visit-to-visit correlation within subjects. The primary test of treatment efficacy was time × treatment interaction. Adjusted changes over time and differences between trial arms were constructed from parameters of the RMANOVA; Test type: Superiority or Other; p = 0.10, RMANOVA — p (within group for subjects receiving norethindrone + conjugated estrogens)=0.05 p (within group for subjects receiving norethindrone + placebo)=0.65 p (between the two groups)=0.10

2. Secondary Outcome: Total Body Bone Mineral Content (BMC)
Time Frame: Baseline to 12 months
Measure: Mean (Standard Error); unit: g
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 25 | 26
g | 37 (10) | 15 (11)
Statistical Analysis 1: Comparison: Intervention Group vs Placebo Group; The time course of each measurement from baseline to 3, 6, 9, and 12 months was compared between arms by repeated-measures analysis of variance (RM-ANOVA), with an autoregressive covariance model to account for visit-to-visit correlation within subjects. The primary test of treatment efficacy was time × treatment interaction. Adjusted changes over time and differences between trial arms were constructed from parameters of the RMANOVA; Test type: Superiority or Other; p = 0.02, RMANOVA — p (within group for participants receiving norethindrone + estrogens)=0.0001 p (within group for participants receiving norethindrone + placebo)=0.31 p (between groups)=0.02

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated every 3 months (at every research visit) for a total of 12 months (the duration of study participation).
Arm/Group | Intervention Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 8/25 | 5/26
Other Adverse Events (participants affected / at risk) | 15/25 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=25) | Placebo Group (N=26)
Hospitalization for pelvic/abdominal pain (Reproductive system and breast disorders) | 3 (4) | 0 (0) — All events determined to be likely due to flare of subject's underlying disease, endometriosis
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 5 (7)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — Bone fractures, secondary to fall or trauma. Non spontaneous, not low impact
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=25) | Placebo Group (N=26)
Myalgias/arthralgias (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 8 (11) | 8 (8) — Pain that did not require hospitalization or surgery
Vaginal bleeding (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Mood swings (Psychiatric disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample of skeletally mature young women; Measurements of aBMD are two-dimensional and do not yield information regarding skeletal strength or microarchitecture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No